CLINICAL TRIAL: NCT03107676
Title: Trunk Extension Endurance Using Four Arms Positions Among Physical Therapy Collegiate Students
Brief Title: Trunk Extension Endurance Among Physical Therapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Collaborators: Cairo University (Other); Taibah University (Other)
Responsible Party: Principal Investigator, Tarek Mohamed El-gohary, Assistant professor doctor, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMR-PT-2017-01
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Spine Injury
Keywords: trunk extensors; endurance, peak torque, power, work
MeSH Terms: conditions — Spinal Injuries

STUDY DESIGN:
Intervention Model Description: Four equal groups of physical therapy students
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessor will only take the endurance and isokinetic measurements without knowing the participants group. Participants will be tested and assigned only to one group using the assigned arms position.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- trunk endurance with hands above head (Active Comparator): participants had to practice trunk extensors endurance training with having hands above head.
  Interventions: Other: trunk extensors endurance training
- trunk endurance with hands behind head (Active Comparator): participants had to practice trunk extensors endurance training with having hands behind head.
  Interventions: Other: trunk extensors endurance training
- trunk endurance with hands parallel (Active Comparator): participants had to practice trunk extensors endurance training with having hands parallel to the trunk.
  Interventions: Other: trunk extensors endurance training
- trunk endurance with no intervention (No Intervention): participants will be tested for trunk extensors endurance with having hands on chest but no intervention.

INTERVENTIONS:
Other: trunk extensors endurance training — endurance training
  Other Names: trunk endurance
  Arms: trunk endurance with hands above head; trunk endurance with hands behind head; trunk endurance with hands parallel

SUMMARY:
College students from physical therapy department will be assigned into four groups. Participants will be tested for trunk extensors endurance and will be given endurance training program to do at home for 6 to 8 weeks. Spinal mobility and lower extremity mobility will be measured. Isokinetic outcome measures for extension and flexion at two different speeds will also be measured at baseline, after 6 and 8 weeks.

DETAILED DESCRIPTION:
Active physical therapy students who are healthy and free from any significant pain at the spine will be recruited to participate in intervention endurance training. Participants will be assigned into four equal groups; doing trunk extension form lying on stomach while breathing normally and arching trunk backwards as long as tolerated. Group one will have arms above head, group two will have hands behind head, group three will have hands parallel to the trunk, and group four will receive instructions only and will act as control group. Spinal mobility of forward bending, backwards bending, right and left side bending will be taken. Straight leg raising and quadriceps flexibility will also be taken. Isokinetic measurements including peak torque, peak torque/body weight, average peak torque, work and average power will be taken at baseline, 6 and 8 weeks. Participants will have a training volume of 2 sets of 10 repetitions, 2 minutes rest in between, 2x/day for 6 to 8 weeks. Endurance timing will be measured in seconds using stop watch. If participant managed to maintain the trunk extension position for 4 minutes, time is recorded and it is considered as ceiling time.

ELIGIBILITY:
Inclusion Criteria:

* Active college student free from any spinal pain or pain 3/10 on pain intensity numeric pain rating scale, willing to participate

Exclusion Criteria:

* have had spinal surgery or pain at the spine more than 3/10 on pain intensity numeric pain rating scale.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
endurance timing | 8 weeks
  trunk extensors endurance timing
isokinetic output | 8 weeks
  peak torque, peak torque/BW, average peak torque, average power, work

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M El-gohary, PhD, Principal Investigator — Taibah University
Locations (1):
- College of Medical Rehabilitation Sciences, Al Madīnah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibrahim Abd Elkader SM, Yehia Al-Shenqiti AM, Fathi El-Gohary TM. Trunk extensors endurance with arms parallel to the trunk is superior to other arms positions: Randomized controlled trial. J Pak Med Assoc. 2022 Feb;72(2):222-227. doi: 10.47391/JPMA.496. PMID 35320165